CLINICAL TRIAL: NCT01299506
Title: An Observational, Multicenter, Open-label Study of the Management of Patients With Advanced Soft Tissue Sarcoma After Failure of Anthracyclines and/or Ifosfamide or Patients Unsuited to Receive These Drugs
Brief Title: Study in Patients With Advanced Soft Tissue Sarcoma (STS) After Failure of Anthracyclines and/or Ifosfamide
Status: Completed | Type: Observational
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: ET-D-010-10
Record Dates: First submitted 2011-02-10; First posted 2011-02-18 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2012-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; trabectedin; Netherlands
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trabectedin: The administration of chemotherapy regimen with trabectedin will be determined by the Investigator's discretion depending on the patients' conditions and previous chemotherapy.
- Conventional care: This includes other palliative chemotherapy or biological therapy or best supportive care.

SUMMARY:
This is an observational, non-randomized, open label, multicenter, phase IV study, which aims to reflect a real-life practice routinely used for the management of advanced soft tissue sarcoma after failure of anthracyclines and/or ifosfamide or patients unsuited to receive these drugs in the Netherlands. This study pretends to reflect the use and schedule of chemotherapy regimen with trabectedin and/or other conventional care regimens such as other palliative chemotherapy/biological therapies or best supportive care (BSC) in the management of advanced soft tissue sarcoma patients in the clinic based at the discretion of the Investigator.

There are no pre-defined limits of administered cycles of trabectedin treatments or chemo- and/or biological therapy; thus, those treatments may continue as long as deemed necessary by the Investigator

DETAILED DESCRIPTION:
* This phase IV study is designed to evaluate, in a real-world setting, usage patterns and associated outcomes associated with the anticancer treatment and/or best supportive care in the clinical practice. The primary study analysis will be to collect clinical data on symptomatic and best response, including tumor control rate, survival, TTP and PFS. Other endpoints of the study will include an evaluation of on-study subsequent anticancer treatments, QoL evaluation by using the EORTC QoL test (QLQ-C30) and an economic cost-effectiveness analysis by using the EQ-5D test.
* The study population will consist of patients with advanced soft tissue sarcoma after failure of anthracyclines and/or ifosfamide or patients unsuited to receive these drugs. To be enrolled in this study, the patients must meet all inclusion criteria and none of the exclusion criteria. Estimated 100 patients will be enrolled.
* Inclusion Criteria

  1. Patients of both sexes with histologically diagnosed advanced soft tissue sarcoma after failure of anthracyclines and/or ifosfamide or patients unsuited to receive these drugs.
  2. Patients must have signed an informed consent document indicating that they understand the purpose and procedures required for the study, and that they are willing to participate in the study.
  3. Age ≥ 18 years. Exclusion Criteria Withdrawal of the informed consent at any point of the study will exclude the patient from the study.
* Assigned Intervention

  1. Trabectedin treatment The administration of chemotherapy regimen with trabectedin will be determined by the Investigator's discretion depending on the patients´ conditions and previous chemotherapy.
  2. Other conventional care regimens: other palliative chemotherapy or biological therapy or best supportive care. Patients on the other conventional care regimens could receive the following preselected treatments options:

A.Palliative chemotherapy or biological therapy (such as Ifosfamide or other anticancer agents with antitumor effect) as a palliative systemic therapeutic modality that may be offered to the patient with advanced soft tissue sarcoma.

B.Best supportive care, as a palliative therapeutic modality that may be offered to the patient with soft tissue sarcoma excluding chemotherapy/biological therapy but including radiotherapy and non-anticancer medication. Hence, this includes nutritional support, analgesics, antibiotics, antiemetic, transfusions, appetitive stimulants, antidepressants or any other symptomatic therapy, palliative surgery and/or psychological support and/or deep relaxation therapy. Localized radiotherapy to alleviate symptoms (i.e., pain) will be allowed, provided that the total delivered dose is within a palliative range. All therapies with potential systemic antitumor effect were excluded as BSC definition

* Subsequent Anticancer Treatments Administered After chemotherapy discontinuation, patients with documented progressive disease (PD) may be treated with subsequent anticancer therapies or best supportive care at the Investigators´ discretion. All subsequent treatments, surgical procedures or radiotherapy will be reported in the CRF.
* The study period starts at study inclusion and will continue until treatment discontinuation, death or until the predefined date of April 2014, when a final analysis have to delivered to the Dutch authorities.
* Efficacy Evaluations: Symptomatic response and best response as per the Investigator, according to RECIST will be assessed. Tumor control rate (CR + PR + SD), TTP, PFS and OS will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with histologically diagnosed advanced soft tissue sarcoma after failure of anthracyclines and/or ifosfamide or patients unsuited to receive these drugs.
* Patients must have signed an informed consent document indicating that they understand the purpose and procedures required for the study, and that they are willing to participate in the study.
* Age ≥ 18 years.

Exclusion Criteria:

* Withdrawal of the informed consent at any point of the study will exclude the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with advanced soft tissue sarcoma after failure of anthracyclines and/or ifosfamide or patients unsuited to receive these drugs. To be enrolled in this study, the patients must meet all inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A J Gelderblom, Prof, Principal Investigator — Leiden University
Locations (5):
- Netherlands (5):
  - NKI Amsterdam, Amsterdam
  - UMC Groningen, Groningen
  - Leiden University, Leiden
  - Nijmegen UMCN, Nijmegen
  - Erasmus MC Rotterdam, Rotterdam